CLINICAL TRIAL: NCT01267942
Title: Single Intraoperative Intravenous Enhancin[Co-amoxiclav] Versus Postoperative Full Oral Course in Prevention of Post Adenotonsillectomy Morbidity:A Randomised Clinical Trial.
Brief Title: Intravenous Enhancin[Co-amoxiclav] Versus Postoperative Enhancin in Prevention of Postadenotonsillectomy Morbidity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nairobi (Other)
Responsible Party: ISSAC MUTHURE MACHARIA/PROFESSOR., University of Nairobi.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P75/4/2008
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2009-10

CONDITIONS: Adenotonsillar Hypertrophy,Under 12 Years.
Keywords: Adenotonsillectomy.
MeSH Terms: interventions — viral enhancing factor, Trichoplusia ni granulosa virus; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous intraoperative Enhancin (Experimental): Patients received a dose of intravenous Enhancin at induction and only oral Paracetamol in the postoperative period.
  Interventions: Drug: Enhancin
- Postoperative oral Enhancin. (Active Comparator): Patients received postoperative oral Enhancin for five days in addition to oral Paracetamol for the same duration. They did not receive an antibiotic during the operation.
  Interventions: Drug: Enhancin

INTERVENTIONS:
Drug: Enhancin — Intravenous Enhancin at induction at a dose of 25 mg/kg amoxycillin equivalent.
  Oral dose of the same at the same dosage for the active comparator arm.
  Other Names: Augmentin.; Clavulin.; Myoclav.; Co- amoxiclav

SUMMARY:
Null hypothesis; The efficacy of Enhancin]Co-Amoxiclav given as a single intravenous dose at induction is not better than a five days oral course of the same given postoperatively in reducing postoperative morbidity after adenotonsillectomy.

DETAILED DESCRIPTION:
Adenotonsillectomy results in morbidity that is reduced by the use of antibiotics.This study had the sole objective of comparing two route of administration to see which has superior results.

ELIGIBILITY:
Inclusion Criteria:

* Patients below 12year scheduled to undergo adenotonsillectomy whose parents or guardians give consent for recruitment into the study.

Exclusion Criteria:

* Non consenting parents or guardians. Antibiotic use in the week preceding surgery. Patients with co mordities. Known allergies to Co-amoxiclav. Patients who develop complication that warrant change of antibiotic.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
POSTOPERATIVE FEVER | OPERATION DAY TO 7 DAYS POSTOPERATIVELY
  Temperature monitored at 1st ,4th and 7th postoperative days.

CONTACTS AND LOCATIONS:
Overall Officials: Musyoka D Mutiso, mmed ent, Principal Investigator — Ministry of Health, Kenya
Locations (1):
- Kenyatta National Hospital., Nairobi, Nairobi County, Kenya

REFERENCES:
- [Background] Colreavy MP, Nanan D, Benamer M, Donnelly M, Blaney AW, O'Dwyer TP, Cafferkey M. Antibiotic prophylaxis post-tonsillectomy: is it of benefit? Int J Pediatr Otorhinolaryngol. 1999 Oct 15;50(1):15-22. doi: 10.1016/s0165-5876(99)00228-1. PMID 10596882
- [Derived] Mutiso MD, Macharia IM. Single intraoperative intravenous Co-Amoxiclav versus postoperative full oral course in prevention of postadenotonsillectomy morbidity: a randomised clinical trial. BMC Ear Nose Throat Disord. 2011 Sep 30;11:9. doi: 10.1186/1472-6815-11-9. PMID 21961644